CLINICAL TRIAL: NCT04784507
Title: En-Bloc Resection of Bladder Tumors: a Multicentric Safety and Feasibility Trial (IDEAL Phase II) vs Conventional Resection of Bladder Tumors?
Brief Title: En-Bloc Resection of Bladder Tumors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Betul Kartal (Other)
Collaborators: Bağcılar Eğitim ve Araştırma Hastanesi (Unknown)
Responsible Party: Sponsor-Investigator, Betul Kartal, Research Coordinator, Medipol University
Organization: Medipol University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 10840098-604.01.01-E.55105
Record Dates: First submitted 2021-02-26; First posted 2021-03-05 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Bladder Neoplasm
Keywords: Urinary Bladder Neoplasms; Urologic Neoplasms; Urogenital Neoplasms
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urologic Neoplasms; Urogenital Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- En Bloc Resection Bladder Tumor (Any energy source) (Experimental): Patients with suspicion of NMIBC (primary or recurrent) that underwent en bloc resection (EBRT
  Interventions: Procedure: En Bloc Resection
- Conventional Transurethral Resection Bladder Tumor (Mono/Bipolar) (Active Comparator): Patients with suspicion of NMIBC (primary or recurrent) that underwent conventional TURBT
  Interventions: Procedure: Conventional Transurethral Resection Bladder Tumor (Mono/Bipolar)

INTERVENTIONS:
Procedure: En Bloc Resection — En bloc transurethral resection of bladder tumor (EBR-BT) using any energy source (laser and bipolar or monopolar energy)
  Arms: En Bloc Resection Bladder Tumor (Any energy source)
Procedure: Conventional Transurethral Resection Bladder Tumor (Mono/Bipolar) — Conventional Transurethral Resection Bladder Tumor (Mono/Bipolar)
  Arms: Conventional Transurethral Resection Bladder Tumor (Mono/Bipolar)

SUMMARY:
Observational data shows that "en bloc" resection of bladder tumor (EBR-BT) may entail advantages when compared with conventional transurethral bladder tumor resection (TURBT). EBR-BT has the potential to increase the rate of correct staging and accurate assignment of risk-classification in non-muscle-invasive bladder cancer (NMIBC) and to avoid re-TURBT in a considerable number of high-grade NMIBC by demonstrating total macro and microscopic eradication of the primary tumor and to provide the basis for a correct treatment based on a correct stage.

Following the rules of the IDEAL collaboration evaluation and stages of surgical innovation and considering EBR-BT as a surgical technical innovation, the investigators designed a multi-institutional, stage 2a/b study on feasibility (procedural success), safety (including pathology features), and short-term efficacy of EBR-BT and as proof of concept on the reliability of NMIBC staging.

Main objective: to prospectively assess the pathological efficacy of EBR-BT in the staging of bladder cancer and the clinical efficacy at short-term recurrence-free survival.

Secondary objectives: To assess the clinical efficacy at short-term (3-months) of EBR-BT, and to compare efficacy in the staging of the EBR-BT with the conventional TURBT.

DETAILED DESCRIPTION:
En-bloc resection of bladder tumors (EBR-BT) has been showing certain advantages over conventional transurethral resection technique (TURBT) in non-muscle-invasive bladder cancer. These advantages consist mainly in the reduction of obturator nerve reflex and obtention of surgical samples according to oncological principles. Advantages in terms of tumor recurrence in the short-term, when compared with TURBT, remain uncertain. Herein several randomized control trials aim to assess comparative outcomes in the short and long term.

A higher rate of detrusor muscle is found in the EBR-BT samples than in the conventional samples resulting in a better staging and at least theoretically the need for fewer re-TURBT indications. However, a detailed and scrupulous description of the histopathological samples is lacking and, it is assumed that the presence of detrusor in the sample without solution of continuity with submucosa and tumor is sufficient to stage. As in surgical samples of other organs, the objective of EBR-RT is not only to obtain detrusor, but also clean margins that ensure the radicality of the tumor.

The hypothesis of the investigators' is that EBR-BT will results in an increased rate of pathological specimen with the presence of detrusor muscle and free-tumor margins, hence a more accurate stage than TURBT and a decrease in 3-months recurrence at short-term (3 months)

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years old and older (adult, older adult) Sexes: All Accepts healthy volunteers: No

Inclusion criteria:

* Patients aged 18 and older presenting with suspicion of primary or recurrent Non-muscle invasive bladder cancer (NMIBC)
* Tumor size estimated by cystoscopy ≤ 3 cm
* Solitary or multiple tumors (up to 3 in number)

Exclusion Criteria:

* Tumor size > 3 cm of maximum dimeter
* Patient with severe systemic disease (ASA III+)
* Location on the anterior bladder wall and/ or anterior bladder neck (relative contraindication depending on accessibility)
* Pregnancy
* Histological diagnosis other than NMIBC urothelial bladder cancer
* Presence or history of previous upper-tract urinary cancer (UTUC)
* Presence of positive cytology without macroscopic identifiable bladder tumor
* Life expectancy < 1 year
* Non-reversible coagulopathy
* Bladder tumor detected during intravesical BCG therapy
* Tumor multiplicity (> 3 tumors)

Contacts and locations:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Pathological Staging | Immediately after the intervention
  Staging of NMIBC is defined by the presence of sufficient detrusor in the EBR-BT specimens, the status of the margins, presence of a tumor and /or CIS in the mucosal margins, the status of the detrusor margin, and suspicion of instability in mucosa free of tumor.
Recurrence at 3 months | 3 months
  Recurrence free survival at 3-months (absence of visible tumors at the site of the previous resection

SECONDARY OUTCOMES:
Operative Complications | intraoperative
  Rate of operative complications (estimated bleeding, bladder perforation, obturatory reflex, tumor fragmentation, conversion to conventional TURBT)
Perioperative Complications | Up to 90 days
  Postoperative complications according to Clavien-Dindo classification

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Bagcilar Education and Research Hospital, Istanbul, Bagcilar
  - Medipol Mega University Hospital, Istanbul, Bagcilar

IPD SHARING:
Plan to Share IPD: Undecided
Data will be provided by request according to the primary objectives of the IPD study and according to the availability in the present trial